CLINICAL TRIAL: NCT07251855
Title: Development and Effectiveness of the Occupational Activities Module on the Quality of Life of Older Persons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Collaborators: Department of Social Welfare, Ministry of Women, Family and Community Development, Malaysia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JEP-2022-677
Record Dates: First submitted 2025-09-29; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Ageing and Geriatric Health
Keywords: Cluster Randomized Trials

STUDY DESIGN:
Intervention Model Description: This study employed a quantitative design using a Cluster Randomized Trial (CRT). This design was chosen because the study involved community centres, the Centre for Older Persons (Pusat Aktiviti Warga Emas, PAWE), making CRT suitable for evaluating new interventions delivered at the organizational or community level. It also helps to prevent contamination between groups, since participants within the same PAWE could otherwise be exposed to both intervention and control activities.
  The study adopted a modified Stepped Wedge approach in the CRT design (SW-CRT). In this modification, only the intervention group implemented the MACK programme in stages, while control group continued usual activities without intervention throughout the study period. This design was considered appropriate because the intervention was expected to be beneficial but could not be delivered to all clusters at the same time due to limitation to the number of assessors and logistics.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention arm received the MACK program, a structured activity-based intervention for older adults delivered over 14 weeks, twice weekly (9:00 a.m.-3:00 p.m.). Sessions were held at PAWE.
  Interventions: Behavioral: Occupational Activities
- Control group (No Intervention): The control group not receiving any intervention. The group continued with PAWE's usual activities that has been established prior to the study.

INTERVENTIONS:
Behavioral: Occupational Activities — The intervention consists of the MACK programme, a structured 14-week activity-based program designed for older adults, delivered twice weekly at PAWE. Unlike general recreational or social programs, MACK provides a standardized framework that combines four domains of engagement such as exercise, sports and games, recreational activities, and social participation. Activities include light to moderate physical exercises, culturally relevant games such as congkak, snakes and ladders, creative tasks like batik painting, and structured group interactions.
  Participants are encouraged to start with light activities and gradually progress in difficulty, with safety measures explained and monitored throughout. Supervisors trained in the MACK module schedule and oversaw activities using a 14-week template to ensure consistency across centers. This distinguishes the intervention from usual PAWE activities, which are unstructured and not guided by a standardized module.
  Arms: Intervention group

SUMMARY:
The purpose of this study was to find out whether the Occupational Activities Module (Modul Aktiviti Cara Kerja - MACK) could help older adults stay more active and healthier. The study examined whether participation in the programme using MACK improved how well older adults carried out their daily activities, how strong and fit they felt, and how good their overall quality of life was.

Two groups of older adults took part. One group joined the MACK programme for 14 weeks, while the other group continued with their normal daily routines. Their ability to perform daily activities, physical fitness, and quality of life were measured at the beginning, middle, and end of the study to identify any changes or improvements.

DETAILED DESCRIPTION:
This study employed a quantitative Cluster Randomized Trial (CRT) design, suitable for community-based settings such as the Centre for Older Persons (Pusat Aktiviti Warga Emas, PAWE), where interventions are delivered at the organizational level. A modified Stepped Wedge CRT (SW-CRT) was used, in which only the intervention clusters implemented the program in a staggered sequence, while control clusters continued routine PAWE activities throughout the study. This design minimized contamination between groups, addressed logistical constraints, and accommodated the limited number of outcome assessors.

The study population consisted of older adults aged 60 years and above who were registered members of PAWE. Most members were local retirees or non-working residents who remained physically and socially active, seeking opportunities to sustain engagement and wellbeing. Sampling was conducted in two stages: (1) selection of PAWE centers and (2) selection of participants within each center. From 28 PAWE centers in the Klang Valley, eight were randomly selected by ballot and then randomly assigned equally to intervention or control groups (n=4 each). Allocation was performed by an independent blinded individual to ensure allocation concealment.

Participant recruitment combined purposive and convenience sampling. PAWE supervisors were briefed on the study and informed eligible members in person or via WhatsApp. The first 10 interested members were listed and screened for eligibility, and seven were selected through simple randomization using Excel's random number generator, with the remaining three held as reserves. The required sample size, calculated using G*Power for repeated-measures ANOVA (α=0.05, power=0.80, effect size=0.19), was 56 participants, adjusted for 10% dropout. Baseline screening used the Modified Barthel Index (MBI) and Mini-Mental State Examination (MMSE).

Inclusion criteria were aged 60 years and above, registered PAWE member, able to communicate in Malay, and not involved in the feasibility study. Exclusion criteria were diagnosis of degenerative disease (e.g., Alzheimer's, Parkinson's, Huntington's, multiple sclerosis), untreatable vision or hearing impairment, moderate to full dependence in ADLs (MBI ≤ 60), or moderate to severe cognitive impairment (MMSE ≤ 20).

The SW-CRT proceeded in four steps. In week 1, all clusters were in control status and baseline assessments were conducted. Beginning in week 2, intervention clusters initiated the program sequentially after baseline assessments, until by week 4 all four intervention PAWE were actively running the program, while control PAWE continued routine activities until the final assessment at week 15. Assessments were conducted at three time points: baseline (P1), mid-intervention at week 8 (P2), and post-intervention at week 15 (P3). Outcome assessors were blinded to allocation status to minimize bias, although participants could not be blinded due to the nature of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years and above.
* Registered member of PAWE.
* Able to understand and communicate in Malay language.
* Not involved in the feasibility study.

Exclusion Criteria:

* Diagnosed with degenerative diseases (e.g., Alzheimer's, Parkinson's, Hungtinton's, multiple sclerosis).
* Untreateable vision or hearing impairment.
* Moderate to full dependence in basic daily activities (MBI score ≤ 60).
* Moderate to severe cognitive impairment (MMSE score ≤ 20).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Modified Barthel Index | Screening of inclusion criteria, Baseline (Before MACK programme), Mid of intervention (Week 8 or after 7 weeks of MACK programme), Post intervention (Week 15 or after 14 weeks of MACK programme
  The Modified Barthel Index (MBI) is a tool to assess functional ability in performing basic activities of daily living (ADL). It evaluates 10 essential activities, including transfers from bed to chair, mobility through walking or wheelchair use, stair climbing, toileting, bladder and bowel control, bathing, dressing, grooming, and feeding. Each activity is scored on a scale from 0 to 10, with the total score ranging from 0 to 100. A total score of 100 indicates full independence, 91-99 reflects minimal assistance, 61-91 indicates moderate assistance, 21-60 reflects substantial assistance, and 0-21 indicates complete dependence in daily functioning. The MBI has demonstrated high internal consistency, with a Cronbach's alpha coefficient of 0.92, confirming its reliability as a measure of functional independence among individuals.
Lawton Instrumental Activities of Daily Living Scale (Lawton IADL) | Baseline (Before MACK programme), Mid of intervention (Week 8 or after 7 weeks of MACK programme), Post intervention (Week 15 or after 14 weeks of MACK programme
  The Lawton Instrumental Activities of Daily Living Scale (Lawton IADL) is used to assess functional ability in performing instrumental activities of daily living, which are more complex than basic daily activities. The instrument evaluates eight domains: ability to use the telephone, shopping, food preparation, housekeeping, laundry, transportation, medication management, and handling finances. Each domain is scored according to the individual's level of independence, with a total score ranging from 0 to 8. A score of 0 indicates low function with dependence on others, while a score of 8 reflects high function and independence. The scale is simple to administer, can be self-reported, and typically takes 10-15 minutes to complete. It has good inter-item reliability (α = 0.85) and demonstrated validity through significant correlations with other functional status measures.
Bruininks Motor Ability Test (BMAT) | Baseline (Before MACK programme), Mid of intervention (Week 8 or after 7 weeks of MACK programme), Post intervention (Week 15 or after 14 weeks of MACK programme
  The Bruininks Motor Ability Test (BMAT) is a standardized assessment used to measure fine and gross motor skills in adults aged 40 years and above. These motor abilities are closely related to physical functioning and the capacity to perform daily activities. The test evaluates performance through subtests and composite structures focusing on fine and gross motor aspects such as balance, mobility, strength, coordination, and object manipulation.
  BMAT comprises comprehensive, stand-alone subtests with established validity, reliability, and sensitivity. Its psychometric properties include test-retest reliability ranging from 0.77 to 0.94, inter-rater reliability between 0.95 and 0.99, and internal consistency values from 0.60 to 0.92. The subtests include fine motor integration, manual dexterity, coordination, balance and mobility, and strength and flexibility.
Older People's Quality of Life Questionnaire - Short Version (OPQOL-Brief) | Baseline (Before MACK programme), Mid of intervention (Week 8 or after 7 weeks of MACK programme), Post intervention (Week 15 or after 14 weeks of MACK programme
  The Older People's Quality of Life Questionnaire Short Version (OPQOL-Brief) is used to assess the quality of life among older adults. Adapted from the original OPQOL with 35 items, the OPQOL-Brief contains 13 items and has been validated in studies conducted in Britain and Italy. It has shown high reliability and validity when compared with other established instruments such as the World Health Organization Quality-of-Life Scale (WHOQOL) and the CASP-19 (Control, Autonomy, Self-Realization, and Pleasure) questionnaire. The internal consistency of the OPQOL-Brief is strong, with a Cronbach's alpha coefficient of 0.856, comparable to that of the original OPQOL.
  Each item is scored on a five-point Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree), with responses reverse-coded for scoring purposes (e.g., 1 = 5, 2 = 4). The maximum possible score is 65, which indicates the highest quality of life, while lower scores reflect poorer quality of life.

OTHER OUTCOMES:
Mini Mental State Examination (MMSE) | Screening of inclusion criteria
  The Mini Mental State Examination (MMSE) is a widely used, simple, and quick tool for assessing cognitive function (Pangman et al., 2000). It evaluates domains such as orientation, registration, attention and calculation, recall, language, and copying. The total score ranges from 0 to 30, with 24-30 indicating no cognitive impairment, 18-23 reflecting mild impairment, and 0-17 suggesting severe impairment. The assessment takes approximately 5-15 minutes to administer. The MMSE demonstrates strong reliability, with Cronbach's alpha coefficients ranging from 0.80 to 0.96.

CONTACTS AND LOCATIONS:
Locations (1):
- Pusat Aktiviti Warga Emas in Klang Valley, Bahagian Warga Emas, Jabatan Kebajikan Masyarakat, Malaysia, Putrajaya, Malaysia

IPD SHARING:
Plan to Share IPD: No